CLINICAL TRIAL: NCT00825253
Title: A Randomised, Open-labelled, 4-period Crossover Trial Characterising Pharmacokinetics and Pharmacodynamics of Biphasic Insulin Aspart 30 Administered Once, Twice or Thrice Daily and Biphasic Human Insulin 30 Administered Once Daily in Subjects With Type 2 Diabetes
Brief Title: Pharmacokinetics and Pharmacodynamics of Biphasic Insulin Aspart 30 and Biphasic Human Insulin 30 in Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1831; 2006-005958-75 (EudraCT Number)
Record Dates: First submitted 2009-01-14; First posted 2009-01-19 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart 30
Drug: biphasic human insulin 30

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to compare the pharmacodynamics (i.e. the glucose-lowering effect of the study medication over the entire observation phase from the time of administration and the efficacy period) and the pharmacokinetics (i.e. amount of the study insulin that can be determined in the blood) of a treatment with biphasic insulin aspart 30 (BiAsp 30) administered once, twice or thrice daily and biphasic human insulin 30 administered once daily in type 2 diabetic subjects

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Type 2 diabetes mellitus diagnosed for at least 12 months prior to screening
* HbA1c value between 7% and 10.5% (both inclusive) at screening
* Any insulin treatment for at least 3 months prior to screening
* Body mass index (BMI): 25 - 40 kg/m2

Exclusion Criteria:

* Use of any oral antidiabetic agent within the past 6 months
* Active proliferative retinopathy or maculopathy requiring treatment within 6 months prior to screening
* Cardiac disease: NYHA class III or IV chronic heart failure (CHF), unstable angina, and/or any myocardial infarction (treated or untreated) within 6 months prior to screening
* Hepatic insufficiency (ALT or AST greater than or equal to 2 times the central laboratory's upper reference limit)
* Renal insufficiency (serum creatinine greater than or equal to 1.6 mg/dL for males; greater than or equal to
* Recurrent hypoglycaemia or hypoglycaemic unawareness
* Anaemia (haemoglobin less than 13.0 mg/dL in males and less than 12.0 mg/dL in females) (WHO criteria)
* Use of any systemic or topical medications (prescribed or non-prescribed) which may alter glucose metabolism (other than insulin products), including but not limited to: systemic or inhaled glucocorticoids, anabolic steroids, non-selective beta-blockers
* History of substance (e.g. drugs, alcohol) abuse or a positive result in the urine drug/alcohol screen or consumption of more than 14 units (women) or 21 units (men) of alcohol per week (One unit of alcohol equals about 250 mL of beer or lager, one glass of wine, or 20 mL spirits)
* Smoking of more than 20 cigarettes per day and inability to refrain from smoking during the in-house period
* Known hepatitis or positive serological tests for the hepatitis B surface antigen (HBsAg) or hepatitis C antibodies or HIV antibodies
* Uncontrolled treated/untreated hypertension (systolic blood pressure greater than or equal to 160 mmHg and/or diastolic blood pressure greater than or equal to 95 mmHg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Heinemann L, Hovelmann U, Brauns B, Nosek L, Haahr HL, Olsen KJ. Biphasic insulin aspart 30/70: pharmacokinetics and pharmacodynamics compared with once-daily biphasic human insulin and Basal-bolus therapy. Diabetes Care. 2009 Aug;32(8):1431-3. doi: 10.2337/dc09-0097. Epub 2009 Jun 1. PMID 19487640
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com